CLINICAL TRIAL: NCT04023552
Title: A Randomized Double-blind, Placebo-controlled, Multicenter Trial Assessing the Impact of Lipoprotein (a) Lowering With Pelacarsen (TQJ230) on Major Cardiovascular Events in Patients With Established Cardiovascular Disease
Brief Title: Assessing the Impact of Lipoprotein (a) Lowering With Pelacarsen (TQJ230) on Major Cardiovascular Events in Patients With CVD
Acronym: Lp(a)HORIZON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTQJ230A12301; CTQJ230A12301 (Other: Novartis); 2019-001076-11 (EudraCT Number)
Expanded Access: NCT07000695 (Available)
Record Dates: First submitted 2019-07-16; First posted 2019-07-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Disease and Lipoprotein(a)
Keywords: Lipoprotein(a),; Lp(a),; CVD,; myocardial infarction,; PAD,; Stroke,; Pelacarsen
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TQJ230 (Experimental): TQJ230 80 mg injected monthly administered subcutaneously
  Interventions: Drug: TQJ230
- Placebo (Placebo Comparator): Monthly subcutaneous injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TQJ230 — TQJ230 80 mg injected monthly administered subcutaneously
  Arms: TQJ230
Drug: Placebo — Placebo to match TQJ230 prefilled syringe to be injected subcutaneously
  Other Names: Placebo to match TQJ230
  Arms: Placebo

SUMMARY:
This is a pivotal phase 3 study designed to support an indication for the reduction of cardiovascular risk in patients with established CVD and elevated Lp(a)

ELIGIBILITY:
Key Inclusion Criteria

* Lp(a) ≥ 70 mg/dL at the screening visit, measured at the Central laboratory
* Myocardial infarction: ≥ 3 months from screening and randomization to ≤ 10 years prior to the screening visit
* Ischemic stroke: ≥ 3 months from screening and randomization to ≤ 10 years prior to the screening visit
* Clinically significant symptomatic peripheral artery disease

Key Exclusion Criteria

* Uncontrolled hypertension
* Heart failure New York Heart Association (NYHA) class IV
* History of malignancy of any organ system
* History of hemorrhagic stroke or other major bleeding
* Platelet count ≤LLN
* Active liver disease or hepatic dysfunction
* Significant kidney disease
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply at the end.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8323 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of clinical endpoint committee confirmed expanded major adverse cardiovascular events in patients with elevated Lp(a) ≥ 70 mg/dL | approximately 4 years
  Demonstrate the superiority of pelacarsen (TQJ230) compared to placebo in reducing the risk of expanded MACE (cardiovascular death, non-fatal MI, non-fatal stroke and urgent coronary re-vascularization requiring hospitalization) in the overall study population with established CVD and (Lp(a) ≥ 70 mg/dL)
Time to the first occurrence of clinical endpoint committee confirmed expanded major adverse cardiovascular events in a population of patients with elevated Lp(a) ≥ 90 mg/dL. | approximately 4 years
  Demonstrate the superiority of pelacarsen (TQJ230) compared to placebo in reducing the risk of expanded MACE (cardiovascular death, non-fatal MI, non-fatal stroke and urgent coronary re-vascularization requiring hospitalization) in the overall study population with established CVD and (Lp(a) ≥ 90 mg/dL)

SECONDARY OUTCOMES:
Time to the first occurrence of the clinical endpoint committee confirmed composite endpoint of major adverse cardiovascular events (CV death, non-fatal MI, and non-fatal stroke) | approximately 4 years
  Demonstrate the superiority of pelacarsen (TQJ230) compared to placebo in reducing the risk of the MACE composite of CV death, nonfatal MI and non-fatal stroke.
Time to the first occurrence of the clinical endpoint committee confirmed composite endpoint of coronary heart disease: coronary heart disease death, non-fatal MI, urgent coronary re-vascularization requiring hospitalization | approximately 4 years
  Demonstrate the superiority of pelacarsen (TQJ230) compared to placebo in reducing the risk of the composite of coronary heart disease (CHD) outcomes: death due to CHD, nonfatal MI and urgent coronary revascularization requiring hospitalization.
Time to Clinical endpoint Committee confirmed all-cause death | approximately 4 years
  Evaluation by clinical endpoint committee the rate of all-cause death
Change in Lp(a) in the log scale from baseline | Baseline, year 1
  Demonstrate the superiority of pelacarsen (TQJ230) compared to placebo in lowering the Lp(a) level at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (758):
- United States (271):
  - SEC Clinical Research LLC, Andalusia, Alabama
  - Grandview Med Group Research LLC, Birmingham, Alabama
  - Novartis Investigative Site, Birmingham, Alabama
  - Heart Center Research Llc, Huntsville, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Mobile Heart Specialists, Mobile, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Cottonwood, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Clinical Research Inst of Arizona, Sun City West, Arizona
  - Novartis Investigative Site, Sun City West, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Cardiology and Medicine Clinic PA, Little Rock, Arkansas
  - Novartis Investigative Site, Little Rock, Arkansas
  - Cardiovascular Res Found, Beverly Hills, California
  - National Heart Institute, Beverly Hills, California
  - Novartis Investigative Site, Beverly Hills, California
  - Flourish Clinical Resrch Covin, Covina, California
  - Novartis Investigative Site, Covina, California
  - Diabetes Lipid Management Center, Huntington Beach, California
  - Novartis Investigative Site, Huntington Beach, California
  - University of Calif Irvine Med Cntr, Irvine, California
  - Novartis Investigative Site, La Jolla, California
  - Memorial Care Health System, Long Beach, California
  - Novartis Investigative Site, Long Beach, California
  - Keck Medical Center USC, Los Angeles, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Novartis Investigative Site, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - University of California San Diego, San Diego, California
  - UCSF, San Francisco, California
  - Novartis Investigative Site, San Francisco, California
  - Helping Hands Medical Associates INC, Santa Ana, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Stanford, California
  - Manshadi Heart Institute, Stockton, California
  - Novartis Investigative Site, Stockton, California
  - Interv Cardiology Med Grp, West Hills, California
  - Novartis Investigative Site, West Hills, California
  - Novartis Investigative Site, Aurora, Colorado
  - Univ Of Color Anschutz Med Center, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Novartis Investigative Site, Bridgeport, Connecticut
  - Novartis Investigative Site, Hartford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Novartis Investigative Site, Boca Raton, Florida
  - Cardiovascular and Vein Center of Florida, Bradenton, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Bay Area Cardiology Assoc., Brandon, Florida
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - CV Consultants of South Broward, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Infinite Clinical Research, Miami, Florida
  - Novartis Investigative Site, Miami, Florida
  - Advanced Research for Health Improvement LLC, Naples, Florida
  - Novartis Investigative Site, Naples, Florida
  - Southwest Florida Research, Naples, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Progressive Medical Research, Port Orange, Florida
  - East Coast Inst for Research LLC, Saint Augustine, Florida
  - Novartis Investigative Site, Saint Augustine, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Novartis Investigative Site, Dunwoody, Georgia
  - Alta Pharmaceutical Research Center, Peachtree Corners, Georgia
  - Cardiovascular Consultants of S GA, Thomasville, Georgia
  - Novartis Investigative Site, Thomasville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Lutheran General Childrens Hospital, Park Ridge, Illinois
  - Novartis Investigative Site, Park Ridge, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Uni Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - University of Kansas Hospital, Kansas City, Kansas
  - Cotton O Neil Clinical Res Center, Topeka, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Christus Health Central Louisiana, Alexandria, Louisiana
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Bogalusa, Louisiana
  - Novartis Investigative Site, Bossier City, Louisiana
  - Cardiovascular Associates Research, Covington, Louisiana
  - Louisiana Heart Center Research, Covington, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Eunice, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Novartis Investigative Site, Hammond, Louisiana
  - CV Institute of the South, Houma, Louisiana
  - Novartis Investigative Site, Houma, Louisiana
  - Horizon Research Grp, Lafayette, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Omega Clinical Research, Metairie, Louisiana
  - Tulane Uni Health Sciences Center, New Orleans, Louisiana
  - Crescent City Physicians Inc, New Orleans, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - CV Ins of the South, Opelousas, Louisiana
  - Novartis Investigative Site, Opelousas, Louisiana
  - Grace Research Llc, Shreveport, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Louisiana Heart Center Research, Slidell, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Zachary, Louisiana
  - Southern Clinical Research, Zachary, Louisiana
  - Maine Health Cardiology, Scarborough, Maine
  - Novartis Investigative Site, Scarborough, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Sinai Ct for Throm Res and Drug Dev, Baltimore, Maryland
  - Johns Hopkins Univ School of Med, Baltimore, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Novartis Investigative Site, Columbia, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Novartis Investigative Site, Ft. Washington, Maryland
  - Adventist HealthCare Shady Grove Medical Center, Rockville, Maryland
  - Novartis Investigative Site, Rockville, Maryland
  - MGH, Boston, Massachusetts
  - Novartis Investigative Site, Boston, Massachusetts
  - Brigham and Womens Hosp Harvard Med School, Boston, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - AA Medical Research Center, Flint, Michigan
  - Novartis Investigative Site, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Novartis Investigative Site, Grand Blanc, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Western Michigan University, Kalamazoo, Michigan
  - McLaren Ctr Research Innovation, Petoskey, Michigan
  - Novartis Investigative Site, Petoskey, Michigan
  - Central Michigan University, Saginaw, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Metro Health Univ of MI Health, Wyoming, Michigan
  - Novartis Investigative Site, Wyoming, Michigan
  - Saint Johns Hospital, Maplewood, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - Belzoni Clinical Research, Belzoni, Mississippi
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Southaven, Mississippi
  - Stern Cardiovascular Foundation Inc, Southaven, Mississippi
  - Novartis Investigative Site, Yazoo City, Mississippi
  - Novartis Investigative Site, City of Saint Peters, Missouri
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Washington Univ School Of Medicine, St Louis, Missouri
  - Mercy South, St Louis, Missouri
  - Mercy Hospital St Louis, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Ridgewood, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Novartis Investigative Site, Summit, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Albany Medical College, Albany, New York
  - Northwell Health, Manhasset, New York
  - Novartis Investigative Site, Manhasset, New York
  - New York Uni Med Ctr, New York, New York
  - Novartis Investigative Site, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Icahn School of Med at Mt Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Northwell Health Physician Peconic, Riverhead, New York
  - Rochester Regional Health, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York
  - Novartis Investigative Site, Southampton, New York
  - Novant Health Heart Vas Inst, Charlotte, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Accellacare US Inc, Raleigh, North Carolina
  - Novartis Investigative Site, Sanford, North Carolina
  - Jones Family Practice PA, Shelby, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Akron Hospital Summa Health System, Akron, Ohio
  - Aultman Hospital, Canton, Ohio
  - Novartis Investigative Site, Canton, Ohio
  - Lindner Ctr At The Christ Hosp, Cincinnati, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Velocity Clin Research Springdale, Cincinnati, Ohio
  - University Of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Rama Research LLC, Marion, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Lancaster General Health, Lancaster, Pennsylvania
  - Novartis Investigative Site, Lancaster, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Novartis Investigative Site, Yardley, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Piedmont Research Partners LLC, Fort Mill, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Germantown, Tennessee
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Apex Cardiology Research Associates of Jackson, Jackson, Tennessee
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Vanderbilt Univ Medi Cen, Nashville, Tennessee
  - Cardiovascular Res of Knoxville LLC, Powell, Tennessee
  - Novartis Investigative Site, Powell, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - SW Family Medicine Associates, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Grace Research, Marshall, Texas
  - Novartis Investigative Site, Temple, Texas
  - Northwest Houston Clinical Research PLLC, Tomball, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Progressive Clinical Research, Bountiful, Utah
  - Intermountain Medical Center, Murray, Utah
  - Novartis Investigative Site, Murray, Utah
  - The University of Utah, Salt Lake City, Utah
  - Novartis Investigative Site, Danville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Novartis Investigative Site, Falls Church, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Novartis Investigative Site, Manassas, Virginia
  - York Clinical Research, Norfolk, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Swedish Medical Center-Cardiovascular Research, Seattle, Washington
  - Univ of Washington Medical Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Novartis Investigative Site, Milwaukee, Wisconsin
  - St Luke s Medical Center Aurora, Milwaukee, Wisconsin
- Argentina (13):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, San Luis
- Australia (7):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Perth, Western Australia
  - Novartis Investigative Site, Liverpool
- Austria (5):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (8):
  - Novartis Investigative Site, Brussels, Brussels Capital
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Aalst, Oost Vlaanderen
  - Novartis Investigative Site, Kortrijk, West-Vlaanderen
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Dendermonde
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Mechelen
- Brazil (19):
  - Novartis Investigative Site, Maceió, Alagoas
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Canoas, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Aracaju, Sergipe
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
- Bulgaria (7):
  - Novartis Investigative Site, Blagoevgrad, Bulgaria
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Pernik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
- Canada (8):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
- Chile (3):
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Santiago
- China (24):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Foshan, Guangdong
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Xiamen
- Colombia (7):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Colombia
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
  - Novartis Investigative Site, San Gil
- Czechia (32):
  - Novartis Investigative Site, Chlumec nad Cidlinou, Chlumec Nad Cidlinou
  - Novartis Investigative Site, Kroměříž, Czech Republic
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Ostrava, Zabreh
  - Novartis Investigative Site, Brandýs nad Labem
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Broumov
  - Novartis Investigative Site, CZE
  - Novartis Investigative Site, Český Krumlov
  - Novartis Investigative Site, Hlučín
  - Novartis Investigative Site, Hodonín
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Liberec
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Mělník
  - Novartis Investigative Site, Most
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Polička
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Přerov
  - Novartis Investigative Site, Slaný
  - Novartis Investigative Site, Svitavy
  - Novartis Investigative Site, Trutnov
  - Novartis Investigative Site, Třebíč
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Valašské Meziříčí
  - Novartis Investigative Site, Zlín
- Denmark (7):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Viborg
- France (11):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valenciennes
- Germany (42):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Künzing, Bavaria
  - Novartis Investigative Site, Muehldorf Am Inn, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Koeln Nippes, North Rhine-Westphalia
  - Novartis Investigative Site, Löhne, North Rhine-Westphalia
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Lutherstadt Witten, Wittenberg
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gelnhausen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Meissen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Saint Ingbert Oberw
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Warendorf
  - Novartis Investigative Site, Weiden
- Greece (5):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chalcis
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Thessaloniki
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, Departamento de Guatemala
  - Novartis Investigative Site, Guatemala City
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Shatin
- Hungary (10):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár
- Iceland (2):
  - Novartis Investigative Site, Kopavogur
  - Novartis Investigative Site, Reykjavik
- India (25):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Guntur, Andhrapradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, Ghaziabad, Uttar Pradesh
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, New Delhi
- Israel (6):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (16):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Napoli
- Japan (33):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Hirosaki, Aomori
  - Novartis Investigative Site, Asahi, Chiba
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Kahoku-gun, Ishikawa-ken
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Komatsu, Ishikawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyhazaki, Miyazaki
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Ōmihachiman, Shiga
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Mexico (5):
  - Novartis Investigative Site, Aguascalientes, Aguascalientes
  - Novartis Investigative Site, Cuernavaca, Morelos
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Culiacan Sinaloa
  - Novartis Investigative Site, Distrito Federal
- Netherlands (24):
  - Novartis Investigative Site, Apeldoorn, Gelderland
  - Novartis Investigative Site, Arnhem, Gelderland
  - Novartis Investigative Site, Nijmegen, Gelderland
  - Novartis Investigative Site, Tiel, Gelderland
  - Novartis Investigative Site, Nijmegen, Gerlderland
  - Novartis Investigative Site, Heerlen, Limburg
  - Novartis Investigative Site, Tilburg, North Brabant
  - Novartis Investigative Site, Alkmaar, North Holland
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Heemstede, North Holland
  - Novartis Investigative Site, Deventer, Overijssel
  - Novartis Investigative Site, Zwolle, Overijssel
  - Novartis Investigative Site, Sneek, Provincie Friesland
  - Novartis Investigative Site, Groningen, Provincie Groningen
  - Novartis Investigative Site, Delft, South Holland
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Leiderdorp, South Holland
  - Novartis Investigative Site, The Hague, South Holland
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Venlo
- Norway (2):
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skedsmokorset
- Novartis Investigative Site, San Miguel, Lima region, Peru
- Poland (10):
  - Novartis Investigative Site, Bielsko-Biala
  - Novartis Investigative Site, Chrzanów
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Kędzierzyn-Koźle
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Sochaczew
  - Novartis Investigative Site, Tarnów
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Setúbal
- Puerto Rico (2):
  - Novartis Investigative Site, Ponce
  - Research and Cardiovascular Corp, Ponce
- Romania (8):
  - Novartis Investigative Site, Buzău, Buzău
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Iași, Jud Iasi
  - Novartis Investigative Site, Baia Mare, Maramureş
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
- Russia (22):
  - Novartis Investigative Site, Saint Petersburg, Russia
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sochy
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Vsevolozhsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (21):
  - Novartis Investigative Site, Brezno, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Dolný Kubín
  - Novartis Investigative Site, Handlová
  - Novartis Investigative Site, Kláštor pod Znievom
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Rimavská Sobota
  - Novartis Investigative Site, Rožňava
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Žilina
- Novartis Investigative Site, Ljubljana, Slovenia
- South Africa (4):
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Cape Town
- South Korea (9):
  - Novartis Investigative Site, Daegu, Dalseo gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Incheon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (16):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Reus, Tarragona
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Huelva
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Switzerland (6):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Liestal
  - Novartis Investigative Site, Zurich
- Taiwan (8):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Hsinchu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
  - Novartis Investigative Site, Yilan
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Ankara, Bilkent-Cankaya
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Samsun, Ilkadim
  - Novartis Investigative Site, Istanbul, Kadikoy
  - Novartis Investigative Site, Eskişehir, Odunpazari
  - Novartis Investigative Site, Samsun, Samsun
  - Novartis Investigative Site, Mersin, Yenisehir
  - Novartis Investigative Site, Izmir
- United Kingdom (39):
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, London, Greater London
  - Novartis Investigative Site, Preston, Lancashire
  - Novartis Investigative Site, Harrow, Middlesex
  - Novartis Investigative Site, Rochdale, North Manchester
  - Novartis Investigative Site, Portadown, Nothern Ireland
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Hardwick, Stockton on Tees
  - Novartis Investigative Site, Chertsey, Surrey
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Sunderland, Tyne and Wear
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, Chichester, West Sussex
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Bromwich
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Londonderry
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Middlesex
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Rhyl
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Swansea
  - Novartis Investigative Site, Tyne and Wear
  - Novartis Investigative Site, Wiltshire
  - Novartis Investigative Site, Wrexham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient -level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with the applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Byambaa E, Roshanravan B, Berglund L. Lipoprotein(a) and CKD: Insights into New Therapeutic Opportunities. Clin J Am Soc Nephrol. 2025 Dec 2. doi: 10.2215/CJN.0000000968. Online ahead of print. PMID 41329869
- [Derived] Cho L, Nicholls SJ, Nordestgaard BG, Landmesser U, Tsimikas S, Blaha MJ, Leitersdorf E, Lincoff AM, Lesogor A, Manning B, Kozlovski P, Cao H, Wang J, Nissen SE. Design and Rationale of Lp(a)HORIZON Trial: Assessing the Effect of Lipoprotein(a) Lowering With Pelacarsen on Major Cardiovascular Events in Patients With CVD and Elevated Lp(a). Am Heart J. 2025 Sep;287:1-9. doi: 10.1016/j.ahj.2025.03.019. Epub 2025 Apr 2. PMID 40185318
- [Derived] Nicholls SJ, Nelson AJ, Michael LF. Oral agents for lowering lipoprotein(a). Curr Opin Lipidol. 2024 Dec 1;35(6):275-280. doi: 10.1097/MOL.0000000000000953. Epub 2024 Sep 25. PMID 39329200
- [Derived] Burvill A, Watts GF, Norman R, Ademi Z. Early health technology assessment of gene silencing therapies for lowering lipoprotein(a) in the secondary prevention of coronary heart disease. J Clin Lipidol. 2024 Nov-Dec;18(6):e946-e956. doi: 10.1016/j.jacl.2024.08.012. Epub 2024 Aug 31. PMID 39322524
- [Derived] Dimitriadis K, Theofilis P, Iliakis P, Pyrpyris N, Dri E, Sakalidis A, Soulaidopoulos S, Tsioufis P, Fragkoulis C, Chrysohoou C, Tsiachris D, Tsioufis K. Management of dyslipidemia in coronary artery disease: the present and the future. Coron Artery Dis. 2024 Sep 1;35(6):516-524. doi: 10.1097/MCA.0000000000001375. Epub 2024 Apr 29. PMID 38682459
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- [Derived] Tsimikas S, Reeves RR, Patel MP. Always Present, But Now Rediscovered: Lp(a) as a Predictor of Long-Term Outcomes in PCI. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2069-2072. doi: 10.1016/j.jcin.2021.08.032. No abstract available. PMID 34556281
- [Derived] Plakogiannis R, Sorbera M, Fischetti B, Chen M. The Role of Antisense Therapies Targeting Lipoprotein(a). J Cardiovasc Pharmacol. 2021 Jul 1;78(1):e5-e11. doi: 10.1097/FJC.0000000000001045. PMID 34232223